CLINICAL TRIAL: NCT02167711
Title: Selective Internal Radiation Therapy With Yttrium-90 Resin Microspheres Followed by Gemcitabine Plus Cisplatin for Intra-hepatic Cholangiocarcinoma: A Phase II Study
Brief Title: Treatment for Bile Duct Cancer in the Liver
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CCTU, Comprehensive Clinical Trial Unit, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTC001
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Cholangio Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SIRT (Experimental)
  Interventions: Drug: SIRT Yttrium-90

INTERVENTIONS:
Drug: SIRT Yttrium-90

SUMMARY:
The current standard treatment of inoperable intrahepatic cholangiocarcinoma (bile duct cancer in the liver) is chemotherapy, which is of limited efficacy. The use of selective internal radiotherapy treatment (SIRT-Y90) is proven efficacious in patients with intra-heptic tumor. Previous experience with SIRT is safe in patients with intrahepatic cholangiocarcinoma. This study aims to study the benefits of sequential administration of SIRT followed by standard chemotherapy for treatment of inoperable intrahepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Histological or cytological diagnosis of cholangiocarcinoma
* Disease not amenable to surgery
* Predominant disease load in the liver (in case of extra-hepatic involvement, only patients with lymph nodes metastases are allowed)
* Naïve to locoregional or systemic treatment (but patients who develop recurrent disease after surgery are suitable)
* ECOG PS 0-1
* At least one measurable disease lesion according to RECIST v 1.1
* Life expectancy of 12 weeks or longer
* Adequate hematological, renal and hepatic function
* Platelet ≥100 x 109
* ANC ≥ 1.5 x 109
* Bilirubin ≤ 30µmol/L
* Albumin ≥ 30g/L
* ALT ≤ 3 ULN
* INR ≤ 1.5
* Serum creatinine ≤ 1.5 x ULN

Exclusion Criteria:

* Prior malignancy except cervical carcinoma-in-situ or treated basal cell carcinoma. Any cancers treated curatively > 5 years prior to study entry are permitted.
* Patients with extra-hepatic disease other than regional lymph node metastases.
* Evidence of ascites or cirrhosis, as determined by clinical or radiologic assessment
* Biliary obstruction with no possibility of drainage
* Non-malignant disease that would render the patient unsuitable for treatment according to the protocol
* Prior treatment of chemotherapy for the cholangiocarcinoma
* Prior radiation therapy to the upper abdomen
* Complete thrombosis of the main portal vein
* Tumor volume > 50% of the normal liver volume
* Allergy to non-ionic contrast agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-09-17 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2 years

SECONDARY OUTCOMES:
Progression-free survival | 2 years
Radiological response | 2 years
disease control rate | 2 years
Duration between timing of chemotherapy and SIRT-Y90 | 2 years
Rate and severity of toxicities | 2 years
Serological response in CA 19.9 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen L Chan, FRCP, Principal Investigator — Department of Clinical Oncology, The Chinese University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong